CLINICAL TRIAL: NCT03205462
Title: An Open Study to Assess the Safety and Pharmacokinetics of Fluorothyazinone Used as a Single-Dose Administration or a Treatment Course in Healthy Volunteers
Brief Title: An Open Study to Assess the Safety and Pharmacokinetics of Fluorothyazinone as a Single-Dose Administration or a Treatment Course in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Collaborators: Center of Pharmaceutical Analytics LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 02-FT-2017
Record Dates: First submitted 2017-06-26; First posted 2017-07-02 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2017-06

CONDITIONS: Healthy Volunteer
Keywords: Pseudomanas Aeruginosa; antibiotic resistance; nosocomial infection; factors of pathogenicity of bacteria; the system of secretion of type III pathogenic bacteria; chronic infection
MeSH Terms: conditions — Cross Infection; Persistent Infection

STUDY DESIGN:
Intervention Model Description: The current Phase I clinical trial has been developed to assess the safety and tolerability of the Fluorothyazinone drug used as a single-dose administration and a treatment course in healthy volunteers. This dose-escalation trial will be conducted with sequential enrollment of volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Fluorothyazinone in a dosage of 300 mg (1 tablet) will be administrated to 5 volunteers
  Interventions: Drug: Fluorothyazinone 300 mg
- Group 2 (Experimental): Fluorothyazinone in a dosage of 600 mg (2 tablets) will be received per os (oral administration) as a single dose
  Interventions: Drug: Fluorothyazinone 600 mg
- Group 3 (Experimental): on the first day of administration, the product is received according to the following regimen: the first dosage of 60 mg (2 tablets) should be taken orally 30 minutes after meals and swallowed with room-temperature water; the second dosage - 1 tablet (300 mg) - 12 hours later, and then for 5 days the subjects will receive 2 tablets per day. The duration of antibacterial therapy is 6 days. The total dose of Fluorothyazinone per treatment course is 3900 mg.
  Interventions: Drug: Fluorothyazinone 3900 mg

INTERVENTIONS:
Drug: Fluorothyazinone 300 mg — Fluorothyazinone in a dosage of 300 mg (1 tablet)
  Arms: Group 1
Drug: Fluorothyazinone 600 mg — Fluorothyazinone in a dosage of 600 mg (2 tablets) is received per os (oral administration) as a single dose
  Arms: Group 2
Drug: Fluorothyazinone 3900 mg — The total dose of Fluorothyazinone per treatment course is 3900 mg.
  Arms: Group 3

SUMMARY:
The current Phase I clinical trial has been developed to assess the safety and tolerability of the Fluorothyazinone drug used as a single-dose administration and a treatment course in healthy volunteers. This dose-escalation trial will be conducted with sequential enrollment of volunteers.

DETAILED DESCRIPTION:
Based on the screening results of volunteers who signed the Informed Consent Form, the volunteers will be sequentially enrolled in three groups to receive different product doses; the total number of volunteers receiving the product will be not less than 25 individuals. In view of the fact that the product will be studied in humans for the first time, initially 5 volunteers will be admitted to the hospital to receive a single product dose. As soon as the product safety is proven by the follow-up period outcomes on Day 7, the study will be continued with the enrollment of additional 5 volunteers. They will receive a single dose of 600 mg to assess the safety and pharmacokinetics of the studied product.

After the interim safety assessment on Day 7 is completed, additional 15 volunteers will enter the study to receive the product in a dosage regimen proposed for the use in clinical practice.

If necessary, backup individuals (not more than 4) will be additionally enrolled in the study. The original volunteers could be replaced only if they had not received the product; in case where a volunteer has received the product, no replacement will take place.

All volunteers will be divided into three groups. Initially, Group I (5 volunteers) will be included in the study. As soon as the interim results of safety tests (complete blood count, clinical biochemical analysis, clinical urine test and clinical examination of the general state of health) obtained on Day 7 are evaluated, the Investigator will make decision on whether to enroll the second group (5 individuals) to assess the product used in a dose of 600 mg. After the interim safety evaluation on Day 7, additional 15 volunteers will enter the study to receive the product in a dosage regimen proposed for use in clinical practice.

Any of the volunteers who received a dose of the studied product will be considered as a subject enrolled in the study, and his/her data will be used for assessing the product safety and tolerability.

The consecutive enrollment of volunteers is implied for each of the groups with an interim assessment of the safety parameters.

The study will be composed of four (4) visits for volunteers of Group I (a screening visit, the hospitalization visit during which a volunteer will receive the studied product and stay for three (3) days at the hospital, and two outpatient visits - 5 and 7 days after receiving the product).

The study will be composed of four (4) visits for volunteers of Group II (a screening visit, the hospitalization visit during which a volunteer will receive the studied product and stay for seven (7) days at the hospital, and two outpatient visits -14 and 28 days after receiving the product).

The study will be composed of five (5) visits for volunteers of Group III (a screening visit, the hospitalization visit during which a volunteer will receive the studied product and stay for seven (7) days at the hospital, and three outpatient visits - 14, 28 and 60 days after receiving the product).

After a volunteer signs the Informed Consent Form at the screening stage, a screening number will be assigned to the volunteer (consecutive numbering system will be used, i.e. numbers will be assigned to volunteers as they arrive: the first volunteer will be assigned a number 01, the second volunteer - 02, the third - 03, etc.), and appropriate notes will be made in the Case Report Forms (CRF) and source documentation.

ELIGIBILITY:
Inclusion Criteria:

* - subject is a male or female between the age of 18 - 45 years;
* subject provides written informed consent;
* subject agrees to use effective contraceptive methods during the entire period of participation in the study (one of the following methods will be used: sexual abstinence; condoms (male or female with or without spermicidal agent); diaphragm or cervical cap with spermicidal agent; intrauterine device); in cases where subjects use hormonal contraceptives, their administration should be discontinued at least 2 months prior to the study commencement date;
* body mass index (BMI) of subject: 18.5 ≤ BMI ≤ 30;
* subject has no acute communicable diseases/recurrence of chronic communicable diseases during the participation in the study and 7 days prior to start of the therapy;
* subject has no severe allergic diseases in the medical history (anaphylactic shock, Quincke's edema, polymorphic exudative eczema, serum disease);
* in medical history and based on the screening results, subject has no diseases of the gastrointestinal system, liver, kidneys, cardiovascular system, CNS, locomotion system, urogenital and endocrine systems that could affect the assessment of the study results;
* subject has a negative result of the blood or urine pregnancy test (for females of childbearing age) not more than 24 hours prior to receiving the first dose of the studied product;
* subject has negative tests for HIV, hepatitis B and c, syphilis;
* subject has a negative result of the urine test for residual narcotic drugs;
* subject has a negative result of the breath alcohol test;
* subject has no hematopoietic malignancies;
* subject has no malignant neoplasms;
* indicators of clinical biochemical analysis, complete blood count and clinical urine test at a screening visit are within the normal range of reference values*

Exclusion Criteria:

* - subject has participated in another clinical trial over the last 90 days;
* subject has experienced symptoms of respiratory disease for the last 3 days;
* subject has received treatment with steroids for the last 10 days (except products for intranasal and topical application);
* subject has received immunoglobulins or other blood products over the last 3 months;
* subject has received immunosuppressive and/or immunomodulating agents within 6 months prior to the start of the study;
* subject has taken medications that have considerable effects on hemodynamics, liver function, etc. (barbiturates, omeprosole, cimetidine, etc.) within less than 30 days prior to the start of the study;
* regular previous or current use of narcotic drugs by subject;
* pregnancy or breast feeding;
* GI system surgeries in subject's history within a one-year period before the subject enters the study;
* subject has systolic blood pressure less than 100 mm Hg or greater than 139 mm Hg; diastolic blood pressure less than 60 mm Hg or greater than 90 mm Hg; heart rate lower than 60 beats per minute or above 90 beats per minute;
* subject has exacerbation of allergic diseases or history of anaphylactic reactions or angioneurotic edema;
* allergic reactions to components of the studied product and concurrent antibacterial agent;
* subject has a concomitant disease which may affect the assessment of the study results: active TB form; chronic hepatic and renal diseases; considerable impairment of thyroid function and other endocrine diseases (diabetes mellitus), severe diseases of the hematopoietic system; epilepsy and other CNS disorders; myocardial infarction in previous history; myocarditis; endocarditis; ischemic heart disease; autoimmune disorders; severe chronic diseases requiring follow-up at the hospital; and, other diseases that, in opinion of the Investigator, will not allow a subject to take part in the study or may affect the study course and/or its results (e.g. assessment of the safety parameters);
* blood donation (at least 450 ml of blood or plasma) by subject in less than 2 months prior to the start of the study;
* subject has a history of the consumption of more than 5 units (0.25 l of pure alcohol) a week
* subject smokes more than 10 cigarettes a day;
* scheduled hospitalization and/or surgery during the period of participation in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Product safety evaluation by assessing its impact on the vital signs (systolic and diastolic blood pressure, heart rate, body temperature) and clinical laboratory test results in healthy volunteers after administration of the product | through study completion, an average of 3 month
  To evaluate the product safety by assessing its impact on the vital signs (systolic and diastolic blood pressure, heart rate, body temperature) and clinical laboratory test results in healthy volunteers after administration of the product

SECONDARY OUTCOMES:
PK parameters: area under the concentration-time curve from time zero to last measurable concentration in blood sample [AUCo-t] | 600 mg - Day 1, Day 2, Day 3; 3900 mg - Day 1, Day 2, Day 3, Day 4, Day 5, Day 6
  To assess the pharmacokinetics in healthy volunteers after the product administration as a single dose of 600 mg (10 time points: Day 1 - prior to the product administration and 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours and 12 hours after the product administration; Day 2 - 24 and 36 hours after the product administration; Day 3 - 48 hours after the product administration) To assess the pharmacokinetics in healthy volunteers after the product administration as dose 3900 mg (18 time points: Day 1 - prior to the product administration and 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours and 12 hours after the product administration; Day 2 - 24 and 36 hours after the product administration; 48 hours after the product administration; Day 4 - 71, 74, 83, 86 hours after the product administration; Day 6 - 119, 122, 131 and 134 hours after the product administration.)
PK parameters: area under the concentration-time curve (from time zero to infinity) [AUCo-∞] | 600 mg - Day 1, Day 2, Day 3; 3900 mg - Day 1, Day 2, Day 3, Day 4, Day 5, Day 6
  To assess the pharmacokinetics in healthy volunteers after product administration as a single dose of 600 mg (10 time points: Day 1 - prior to the product administration and 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours and 12 hours after the product administration; Day 2 - 24 and 36 hours after the product administration; Day 3 - 48 hours after the product administration) To assess the pharmacokinetics in healthy volunteers after the product administration as dose 3900 mg (18 time points: Day 1 - prior to the product administration and 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours and 12 hours after the product administration; Day 2 - 24 and 36 hours after the product administration; 48 hours after the product administration; Day 4 - 71, 74, 83, 86 hours after the product administration; Day 6 - 119, 122, 131 and 134 hours after the product administration.)
PK parameters: the maximum concentration [Cmax] | 600 mg - Day 1, Day 2, Day 3; 3900 mg - Day 1, Day 2, Day 3, Day 4, Day 5, Day 6
  To assess the pharmacokinetics in healthy volunteers after product administration as a single dose of 600 mg (10 time points: Day 1 - prior to the product administration and 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours and 12 hours after the product administration; Day 2 - 24 and 36 hours after the product administration; Day 3 - 48 hours after the product administration) To assess the pharmacokinetics in healthy volunteers after the product administration as dose 3900 mg (18 time points: Day 1 - prior to the product administration and 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours and 12 hours after the product administration; Day 2 - 24 and 36 hours after the product administration; 48 hours after the product administration; Day 4 - 71, 74, 83, 86 hours after the product administration; Day 6 - 119, 122, 131 and 134 hours after the product administration.)
PK parameters: time to reach the maximum concentration [Tmax] | 600 mg - Day 1, Day 2, Day 3; 3900 mg - Day 1, Day 2, Day 3, Day 4, Day 5, Day 6
  To assess the pharmacokinetics in healthy volunteers after product administration as a single dose of 600 mg (10 time points: Day 1 - prior to the product administration and 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours and 12 hours after the product administration; Day 2 - 24 and 36 hours after the product administration; Day 3 - 48 hours after the product administration) To assess the pharmacokinetics in healthy volunteers after the product administration as dose 3900 mg (18 time points: Day 1 - prior to the product administration and 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours and 12 hours after the product administration; Day 2 - 24 and 36 hours after the product administration; 48 hours after the product administration; Day 4 - 71, 74, 83, 86 hours after the product administration; Day 6 - 119, 122, 131 and 134 hours after the product administration.)
PK parameters: half-life [T1/2] | 600 mg - Day 1, Day 2, Day 3; 3900 mg - Day 1, Day 2, Day 3, Day 4, Day 5, Day 6
  To assess the pharmacokinetics in healthy volunteers after product administration as a single dose of 600 mg (10 time points: Day 1 - prior to the product administration and 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours and 12 hours after the product administration; Day 2 - 24 and 36 hours after the product administration; Day 3 - 48 hours after the product administration) To assess the pharmacokinetics in healthy volunteers after the product administration as dose 3900 mg (18 time points: Day 1 - prior to the product administration and 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours and 12 hours after the product administration; Day 2 - 24 and 36 hours after the product administration; 48 hours after the product administration; Day 4 - 71, 74, 83, 86 hours after the product administration; Day 6 - 119, 122, 131 and 134 hours after the product administration.)
PK parameters: elimination rate constant [kel] | 600 mg - Day 1, Day 2, Day 3; 3900 mg - Day 1, Day 2, Day 3, Day 4, Day 5, Day 6
  To assess the pharmacokinetics in healthy volunteers after product administration as a single dose of 600 mg (10 time points: Day 1 - prior to the product administration and 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours and 12 hours after the product administration; Day 2 - 24 and 36 hours after the product administration; Day 3 - 48 hours after the product administration) To assess the pharmacokinetics in healthy volunteers after the product administration as dose 3900 mg (18 time points: Day 1 - prior to the product administration and 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours and 12 hours after the product administration; Day 2 - 24 and 36 hours after the product administration; 48 hours after the product administration; Day 4 - 71, 74, 83, 86 hours after the product administration; Day 6 - 119, 122, 131 and 134 hours after the product administration.)
PK parameters: volume of distribution [Vd] | 600 mg - Day 1, Day 2, Day 3; 3900 mg - Day 1, Day 2, Day 3, Day 4,Day 5, Day 6
  To assess the pharmacokinetics in healthy volunteers after product administration as a single dose of 600 mg (10 time points: Day 1 - prior to the product administration and 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours and 12 hours after the product administratio; Day 2 - 24 and 36 hours after the product administration; Day 3 - 48 hours after the product administration) To assess the pharmacokinetics in healthy volunteers after the product administration as dose 3900 mg (18 time points: Day 1 - prior to the product administration and 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours and 12 hours after the product administration; Day 2 - 24 and 36 hours after the product administration; 48 hours after the product administration; Day 4 - 71, 74, 83, 86 hours after the product administration; Day 6 - 119, 122, 131 and 134 hours after the product administration.)
PK parameters: relative rate of absorption [Cmax/AUC] | 600 mg - Day 1, Day 2, Day 3; 3900 mg - Day 1, Day 2, Day 3, Day 4, Day 5, Day 6
  To assess the pharmacokinetics in healthy volunteers after product administration as a single dose of 600 mg (10 time points: Day 1 - prior to the product administration and 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours and 12 hours after the product administration; Day 2 - 24 and 36 hours after the product administration; Day 3 - 48 hours after the product administration) To assess the pharmacokinetics in healthy volunteers after the product administration as dose 3900 mg (18 time points: Day 1 - prior to the product administration and 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours and 12 hours after the product administration; Day 2 - 24 and 36 hours after the product administration; 48 hours after the product administration; Day 4 - 71, 74, 83, 86 hours after the product administration; Day 6 - 119, 122, 131 and 134 hours after the product administration.)

CONTACTS AND LOCATIONS:
Locations (1):
- Federal State Budget-Funded Educational Institution for Additional Professional Education "Russian Medical Academy for Postgraduate Education" of the Ministry of Health of the Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided